CLINICAL TRIAL: NCT03293069
Title: Conservative Iron Chelation as a Disease-modifying Strategy in Amyotrophic Lateral Sclerosis: Multicentre, Parallel-group, Placebo-controlled, Randomized Clinical Trial of Deferiprone
Brief Title: Conservative Iron Chelation as a Disease-modifying Strategy in Amyotrophic Lateral Sclerosis
Acronym: FAIR-ALS II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016_76; 2017-003763-35 (EudraCT Number)
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Conservative Iron Chelation; Disease-modifying Strategy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Deferiprone; Isoflurophate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deferiprone (Experimental): Half of participants will receive twice-daily oral deferiprone taken over 12 months.
  Interventions: Drug: Deferiprone
- Placebo (Placebo Comparator): Half of participants will receive the placebo Twice-daily oral placebo taken over 12 months
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Deferiprone — One 600 mg delayed-release tablets of deferiprone twice a day, for at 30 mg/kg/day
  Other Names: DFP
  Arms: Deferiprone
Drug: Placebo Oral Tablet — the placebo twice daily morning and evening.
  Arms: Placebo

SUMMARY:
The alteration of iron metabolism is reported in animal models of amyotrophic lateral sclerosis (ALS) as well as in sporadic and genetic forms (SOD1 and C9orf72) of ALS. The high iron concentration of the brain, due to its high energy demand (high oxygen consumption), makes motor neurons particularly vulnerable to energy deficit and oxidative stress. Post-mortem examinations and MRI scans in patients with ALS have found signs of iron accumulation in the central motor tract; and a high level of serum ferritin, which is a marker of iron levels, is associated with a lower prognosis. In ALS mouse models, the use of iron chelators has demonstrated neuroprotection and increased life expectancy, suggesting that elimination of excess iron from the brain can prevent neuronal loss and, consequently, a slow progression of the disease. Conservative chelation of iron refers to a modality whereby much of the iron that binds to the chelator is redistributed in the body rather than exhausted. Using a chelator, deferiprone, with this feature, in a safety pilot study, a very good safety profile was observed. Deferiprone eliminated excess iron from brain regions, reduced oxidative damage and cell death associated with regional iron deposits with no apparent negative impact on the iron levels needed. Now, the efficacy of this new therapeutic modality of neuroprotection is being evaluated in a randomized, double-blind, placebo-controlled, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Categorized as; possible, laboratory supported probable, probable, or definite ALS (revised El Escorial criteria)
* Spinal and bulbar forms of ALS
* Duration of the disease of less than 18 months since the first symptoms of motor deficit or amyotrophy (isolated cramps or fasciculation will not be considered).
* Duration of the disease of less than 6 months since the diagnosis
* An upright slow vital capacity ≥ 75% of the predicted value for age, height, and sex or at least one test on inspiratory pressure ≥ 60% of the predicted value for age, height, and sex which could be either maximal inspiratory pressure or a SNIFF test. (The best predictive test is sniff test but sometime patients are not able to do it.) (In case of a limit abnormal value for one of them, it will be recommended that patient re-assessment occurs three months later).
* A mild functional handicap score for ALSFRS-R ≥36
* An upright slow vital capacity > 70% of the predicted value for age, height, and sex and
* Able to swallow (required for oral treatment)
* Patients weight included between 40 kg and 130 kg
* If the patient is under riluzole, it has to be for at least 1 month before inclusion with stable dose (to rule out the principal risk of hepatitis)

Exclusion Criteria:

* Patients with high frequency of comorbidity or vital risks that may reasonably impair life expectancy
* Progressing axis I psychiatric disorders (psychosis, hallucinations, substance addiction, bipolar disorder, severe depression, suicidal ideation), in accordance with the Diagnostic and Statistical Manual of Mental Disorders. Before entry into the study, exclusion or stabilization of conditions must occur for patients suffering from mild or moderate depressive episodes (not in remission) or severe and uncontrolled anxiety.
* Dementia according to the Diagnostic and Statistical Manual of Mental Disorders
* Exposure to any other experimental drug up to 30 days before day 1
* Due to the risk of agranulocytosis (estimated at 2%) caused by the Investigational Medicinal Products (IMPs) and the unknown mechanism by which this agranulocytosis is induced, combining Deferiprone with other medicinal products known to cause agranulocytosis (as described in the IB) will not be allowed. Such medicinal products include clozapine as well as some NSAIDs (e.g. Phenylbutazone or Metamizole), antithyroid agents, sulfonamide antibiotics or methotrexate.
* A history of relapsing neutropenia
* Patients with agranulocytosis or with a history of agranulocytosis.
* Hypersensitivity to Deferiprone
* Patients with anaemia (regardless of latter aetiology) or a history of another haematological disease. Haemochromatosis is not an exclusion criterion if controlled.
* Pregnant or breastfeeding women or women of childbearing potential not taking highly effective contraception.
* Kidney or liver failure.
* Inability to provide informed consent.
* Participation in another clinical trial within 1 month prior to inclusion in the study
* Patients under trusteeship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
CAFS score (Combined Assessment of Function and Survival) | at 12 months
  CAFS score based on changes in amyotrophic lateral sclerosis functional rating scale (ALSFRS-R) total scores and time to death from baseline (randomization visit) to 12 months

SECONDARY OUTCOMES:
Changes in ALS Functional Rating Scale-Revised (ALSFRS-R) total score | Baseline, at 12 months
All-cause and respiratory insufficiency mortality | at 12 months
  Time to death for all cause or respiratory insufficiency (defined as tracheostomy or the use of non-invasive ventilation for ≥ 23 h per day for 14 consecutive days) from baseline until 12 month
Changes in muscle strength | Baseline, at 12 months
  Muscle strength measurements are determined by the overall mega-score for handheld dynamometry and manual muscular testing with a validated medical device provided
Change in the slow vital capacity | Baseline, at 12 months
  The slow vital capacity is measure by the maximum amount of air that can be exhaled following a deep breath. Reflecting the Respiratory insufficiency.
Changes in body weight | Baseline, at 12 months
Change in Quality of life | Baseline, at 12 months
  Quality of life assessed using the five-item form of the ALS assessment questionnaire (ALSAQ-5) from baseline to 12 months
DSMIV criteria | at 12 months
  Dementia (yes/no)
Fronto-Temporal Dementia (FTD) criteria | at 12 months
  Using the revised guidelines for the diagnosis of behavioral variant frontotemporal dementia based on recent literature and collective experience by Rascovsky K et al 2011; Lamarre AK et al 2013
Change in Montreal Cognitive Assessment (MoCA) | Baseline, at 12 months
  MoCA evaluated of mild cognitive dysfunction.
Change in Edinburgh Cognitive and Behavioural Amyotrophic Lateral Sclerosis Screen (ECAS) | Baseline, at 12 months
  ECAS determine cognitive and behavioral changes of patients suffering from Amyotrophic Lateral Sclerosis.
  With ECAS, ALS-specific (fluency, executive functions and social cognition, language) and ALS-nonspecific (memory, visuospatial functions) functions can be analyzed to enable the distinction from other diseases with cognitive and behavioral impairments.

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (15):
- France (15):
  - Chr Angers, Angers
  - Chru Brest, Brest
  - Hopital Pierre Wertheimer - Hcl - Bron, Bron
  - Chu Cote de Nacre - Caen, Caen
  - Chu de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Roger Salengro, CHU, Lille
  - C H U Dupuytren Limoges, Limoges
  - Aphm Hopital La Timone, Marseille
  - Chu de Nancy, Nancy
  - Chu de Nice Hopital Pasteur, Nice
  - Hu Pitie Salpetriere Aphp, Paris
  - Hopital de Hautepierre, Strasbourg
  - Chu de Bordeaux - Talence, Talence
  - Chu Toulouse, Toulouse
  - Chu de Tours, Tours